CLINICAL TRIAL: NCT06947057
Title: Classifying Fully Guided Surgical Guides: A Comprehensive Analysis of Accuracy
Brief Title: Classifying Fully Guided Surgical Guides
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111333
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dental Prostheses
Keywords: Guided implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unilateral tooth supported (Active Comparator): Unilateral guided implant placement
  Interventions: Procedure: Guided implant placement
- Bilateral tooth supported (Active Comparator): Bilateral guided implant placement
  Interventions: Procedure: Guided implant placement
- Full arch mucosa supported (Active Comparator): Full arch implant placement mucosa supported
  Interventions: Procedure: Guided implant placement
- Stackable bone supported (Active Comparator): Stackable guide, foundation guide and on top implant placement guide
  Interventions: Procedure: Guided implant placement

INTERVENTIONS:
Procedure: Guided implant placement — The four types of fully guided surgical guides (bilateral tooth-supported guides, unilateral tooth-supported guides, mucosa-supported full arch guides and stackable guides)

SUMMARY:
Surgical guides can be classified according to support into tooth-supported, mucosa-supported, bone-supported, or a combination of these. Tooth-supported templates are further divided into unilateral or bilateral tooth support. Bilateral tooth-supported guides refer to templates that are supported by templates on both sides while unilateral tooth support refers to templates that is supported by teeth on one side and mucosa or bone from the other side. Usually, mucosa-supported guides are utilized in full arch cases in which there is no need for bone reduction. Stackable guides are the best option when bone reduction is indicated because they allow for the planning of both implant osteotomies and bone sculpturing using a single template made up of different components. This study compare all static guided protocols( bilateral tooth supported, unilateral tooth supported, full arch mucosa supported, stackable bone supported ) with each other under homogenous conditions.

DETAILED DESCRIPTION:
Surgical guides can be classified according to support into tooth-supported, mucosa-supported, bone-supported, or a combination of these. Tooth-supported templates are further divided into unilateral or bilateral tooth support. Bilateral tooth-supported guides refer to templates that are supported by templates on both sides while unilateral tooth support refers to templates that is supported by teeth on one side and mucosa or bone from the other side. Usually, mucosa-supported guides are utilized in full arch cases in which there is no need for bone reduction. Stackable guides are the best option when bone reduction is indicated because they allow for the planning of both implant osteotomies and bone sculpturing using a single template made up of different components.

Theoretically, bilateral tooth-supported guides offer the most accuracy since they offer the best retention and biomechanical stability with anchorage on hard tissues. According to a recent systematic review, unilateral tooth guides exhibited higher deviations except in global coronal deviation where unilateral tooth-supported guides exhibited slightly lower distribution than bilateral guides, and in in vivo global apical deviation where bilateral and unilateral tooth-supported guides showed a similar data range.

Despite the increasing predictability of guided surgery, there will always be differences between the virtual plan and actual performance. The accuracy of static computer-aided implant operations was assessed in the 2018 International Team for Implantology consensus document. According to the study, the variations for the mean crestal point, apical point, angle, coronal depth, and apical depth were 1.2 mm, 1.4 mm, 3.5 o, 0.2 mm, and 0.5 mm, respectively. A safety margin of 2 mm ought to be taken into account at all times, based on the previously indicated precision.

For the purposes of this study, accuracy is defined as the closeness of spatial agreement between any given implant as planned (reference) and as inserted (measurement), expressed by four spatial deviation parameters

ELIGIBILITY:
Inclusion Criteria:

* Missing either only one tooth or partially or fully edentulous.
* Good oral hygiene.
* Systemic free.

Exclusion Criteria:

* Conditions that might render intraoral manipulation impossible (limited mouth opening, excessive gag reflex).
* Bisphosphonate treatment (either at the time of screening or in the history).
* Radiotherapy, irradiation of the mandible or the maxilla (either at the time of screening or in the history).
* Smokers.
* Untreated periodontal disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Angular deviation | Immediately postoperative
  The angle closed by the principal axis of the planned implant and the principal axis of the inserted implant in degrees